CLINICAL TRIAL: NCT00469183
Title: An Assessment of the Atrophogenic Potential of Triple Combination Cream Using Histology Measures in the Treatment of Moderate to Severe Melasma
Brief Title: Assessment of Atrophogenic Potential of Triple Combination Cream for Treatment of Melasma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Ronald W. Gottschalk, MD / Medical Director, Galderma laboratories, L.P.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: US10010
Record Dates: First submitted 2007-05-02; First posted 2007-05-04 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2008-03

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis | interventions — Fluocinolone Acetonide; hydroquinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Fluocinolone acetonide .1%, hydroquinone 4%, tretinoin .05% — Apply topically daily for 12 weeks and continue until condition is clear or almost clear for up to 24 weeks; Maintenance phase: Apply topically twice weekly until the end of study (24 weeks) or condition relapses
  Other Names: TriLuma Cream

SUMMARY:
Evaluate atrophogenic potential of long-term use of Tri-Luma Cream on facial Melasma through biopsy examination.

DETAILED DESCRIPTION:
Same as above.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a clinical diagnosis of moderate to severe melasma
* Subjects willing to undergo biopsy four times throughout the study, two biopsies at baseline (one in a melasma involved area and one in a non-involved area). The third and fourth biopsies will be performed at 3 months and 6 months, respectively; in order to avoid variability in histopathological findings,
* Subjects must have substantial melasma involvement of the cheeks and be willing to have the same general site biopsied at the baseline, month 3 and month 6 visits.

Exclusion Criteria:

* Subjects with diagnosis of dermal melasma
* Subjects who foresee intensive UV exposure during the study (mountain sports, UV radiation, sunbathing, etc.)
* Subjects who have used retinoids, steroids, and/or skin lightening products 4 weeks prior to study entry
* Subjects who show signs of Poikiloderma of Civatte (mandibular hyperpigmentation)
* Subjects with a history of hypertrophic scarring or a history of keloids
* Subjects who are unable to avoid the use of a class 1 steroid during their participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-05; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Safety - Skin biopsy evaluation - histological assessment of skin atrophy | Baseline, 12 weeks and 24 weeks

SECONDARY OUTCOMES:
Tolerability assessments; Incidence of adverse events; Global Assessment of Lesion Severity; MASI; Physician Global Assessment | Baseline, 12 weeks and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ronald W Gottschalk, MD, Study Director — Galderma R&D
Locations (2):
- United States (2):
  - Vitiligo and Pigmentation Institute of Southern California, Los Angeles, California
  - University of Texas Southwestern Medical Center of Dallas, Dallas, Texas

REFERENCES:
- [Derived] Grimes PE, Bhawan J, Guevara IL, Colon LE, Johnson LA, Gottschalk RW, Pandya AG. Continuous therapy followed by a maintenance therapy regimen with a triple combination cream for melasma. J Am Acad Dermatol. 2010 Jun;62(6):962-7. doi: 10.1016/j.jaad.2009.06.067. Epub 2010 Apr 15. PMID 20398959